CLINICAL TRIAL: NCT04407741
Title: An Open-Label Phase Ⅰ/Ⅱ Study of EZH2 Inhibitor SHR2554 in Combination With Anti-PD-L1/TGFβ Antibody SHR1701 in Patients With Advanced or Metastatic Solid Tumors and Relapsed/Refractory B-cell Lymphomas
Brief Title: Phase Ⅰ/Ⅱ Study of SHR2554 in Combination With SHR1701 in Patients With Advanced Solid Tumors and B-cell Lymphomas
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Bio-therapeutic Department, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-055
Record Dates: First submitted 2020-05-20; First posted 2020-05-29 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Solid Tumor; Lymphoma
Keywords: Anti-PD-L1/TGFβ; EZH2; SHR2554; SHR1701; Advanced
MeSH Terms: conditions — Lymphoma | interventions — SHR-1701

STUDY DESIGN:
Intervention Model Description: In phase I period, patients that meet inclusion and exclusion criteria are enrolled to evaluate the safety, feasibility and pharmacokinetics of SHR2554 plus SHR1701. In the following phase II period, based on the recommended dose level from phase I study, enrolled patients are randomized to trial group (SHR2554 plus SHR1701) and control group (SHR1701) to assess the clinical efficacy of SHR2554 plus SHR1701 and immunomodulating effect of SHR2554 to SHR1701 in each cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR2554+ SHR1701 (Experimental): Drug: SHR2554 recommended dose from phase Ⅰstudy, PO, twice a day, every 3 weeks SHR1701 30mg/kg IV over 30 minutes on day 1, every 3 weeks
  Interventions: Drug: SHR2554+SHR1701
- SHR1701 (Experimental): Drug: SHR1701 30mg/kg IV over 30 minutes on day 1, every 3 weeks
  Interventions: Drug: SHR1701

INTERVENTIONS:
Drug: SHR2554+SHR1701 — SHR2554: recommended dose from phase I trial, PO, twice a day. SHR1701: 30mg/kg, IV, over 30 minutes
  Arms: SHR2554+ SHR1701
Drug: SHR1701 — SHR1701: 30mg/kg, IV, over 30 minutes
  Arms: SHR1701

SUMMARY:
The potency of immune checkpoint blockade is limited in most solid malignancies, one possible reason for which is tumor microenvironment. Enhancer of zeste homolog 2 (EZH2) as a epigenetic target for cancer therapy has attracted significant interest. The combination of EZH2 inhibitors and programmed death-1 ligands/ transforming growth factor-β (PD-L1/TGFβ) blockade may enhance the efficiency of immunotherapy.The primary objective of this study in phase Ⅰstage is to assess the safety, feasibility of EZH2 inhibitor SHR2554 in combination with anti-PD-L1/TGFβ antibody SHR1701 in advanced pretreated solid tumors and b-cell lymphomas. The phase Ⅱ stage of this study is to primarily evaluate the efficacy of SHR2554 plus SHR1701 and the epigenetic modulating effect of SHR2554.

DETAILED DESCRIPTION:
Immune checkpoint blockade has led to great strides in the management of various cancers, however, durable response could be seen in approximately 20% of treated patients with most solid malignancies. Immunosuppressive entities such as transforming growth factor-β (TGF-β) in the tumor microenvironment (TME) remain a major impediment. Enhancer of zeste homolog 2 (EZH2) is the core component of the polycomb group complex, which play a major role in cellular proliferation and differentiation. EZH2 aberration has been seen in a wide range of solid tumors and hematological malignancies, affecting tumor progression and immune cells in the tumor microenvironment, and it is associated with poor clinical prognosis and outcomes. EZH2 is not only an activator of gene expression through different pathways, but also a critical epigenetic repressor through histone methylation. Therefore, EZH2 has attracted significant interest as a potential epigenetic target for cancer treatment. It is hypothesized that the combination of EZH2 inhibitors and programmed death-1 ligands/ transforming growth factor-β (PD-L1/TGFβ) blockade could enhance the efficiency of immunotherapy.

The primary objective of this study in phase Ⅰstage is to assess the safety, feasibility of EZH2 inhibitor SHR2554 in combination with anti-PD-L1/TGFβ antibody SHR1701 in advanced pretreated solid tumors and b-cell lymphomas. The second objectives include characterizing the pharmacokinetics of SHR2554 in combination with SHR1701, evaluating the preliminary efficacy of SHR2554 plus SHR1701 and the epigenetic modulating effect of SHR2554 in its combination with anti-PD-L1/TGFβ antibody. The exploratory objectives are to evaluate the pathological, immunological or clinical predictive factors for efficacy and toxicity. Based on the data of safety, efficacy and recommended dose level obtained from phase Ⅰtrial, this study moves into phase Ⅱ stage, in which enrolled subjects are randomized to SHR2554 plus SHR 1701 or SHR1701 monotherapy, to primarily evaluate the efficacy of SHR2554 plus SHR1701 and the epigenetic modulating effect of SHR2554. The second objectives include evaluating safety and other efficacy parameters, such as overall response rate (ORR), disease control rate (DCR), duration of response (DOR) and overall survival (OS). The exploratory objectives are to evaluate laboratory predicting biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age from 18 to 70 years with estimated life expectancy >3 months.
* 2. Histopathological confirmed locally advanced or metastatic systematically pretreated epidermal growth factor receptor (EGFR) / anaplastic lymphoma kinase (ALK) / c-ros oncogene 1 receptor kinase (ROS1) /BRAF negative non-small cell lung cancer (adenocarcinoma or squamous cell carcinoma), pancreatic adenocarcinoma, cholangiocarcinoma, gastrointestinal adenocarcinoma, triple-negative breast cancer and relapsed/refractory B-cell lymphoma (All enrolled subjects with above solid carcinoma are required to have received at least first-line systematic therapy and subjects with R/R B-cell lymphoma need a history of at least two lines of previous treatment; For solid carcinoma subjects enrolled in phase Ⅱ period, their previous treatment lines are limited to no more than four lines; Besides previously treated subjects, subjects with initially diagnosed pancreatic adenocarcinoma or cholangiocarcinoma are also eligible for enrollment in phase Ⅱ period).
* 3. Have at least one measurable target lesion, determined by the site study team based on RECIST 1.1 and immune related RECIST.
* 4. Fresh tumor samples or formalin-fixed paraffin embedded tumor archival samples within 3 months are necessary; Fresh tumor samples are preferred. Subjects are willing to accept tumor re-biopsy in the process of this study.
* 5. Previous treatment must be completed for more than 4 weeks prior to the enrollment of this study, and subjects have recovered to <= grade 1 toxicity.
* 6. Have an Eastern Cooperative Oncology Group performance status (ECOG) of 0 or 1 at the time of enrollment.
* 7. Have adequate organ function, as defined in the table below, which should be confirmed within 2 weeks prior to the first dose of study drugs.

  * Leukocytes greater than or equal to 3.0 ×10^9/L.
  * Absolute neutrophil counts greater than or equal to 1.0 ×10^9/L.
  * Platelets greater than or equal to 100 ×10^9/L.
  * Hemoglobin greater than or equal to 90 g/L.
  * Total bilirubin less than or equal to 2 x ULN.
  * Serum albumin should be no less than 30 g/L.
  * Alanine aminotransferase or Aspartate aminotransferase less than 2 x Upper Limit of Normal (ULN).
  * Measured creatinine clearance ≥ 60 mL per min.
* 8. Previous treatment with anti-PD-1/PD-L1 antibodies or cytotoxic T lymphocyte associated antigen 4 (CTLA-4) inhibitors are allowed.
* 9. Ability to understand and sign a written informed consent document.
* 10.Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, and up to 90 days after the last dose of the drug.

Exclusion Criteria:

* 1. Active, known or suspected autoimmune diseases.
* 2. Known brain metastases or active central nervous system (CNS). Subjects with CNS metastases who were treated with radiotherapy for at least 3 months prior to enrollment, have no central nervous symptoms and are off corticosteroids, are eligible for enrollment, but require a brain MRI screening.
* 3. Subjects are being treated with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment.
* 4. History of severe hypersensitive reactions to other monoclonal antibodies.
* 5. History of allergy or intolerance to study drug components.
* 6. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
* 7. History or concurrent condition of interstitial lung disease of any grade or severely impaired pulmonary function.
* 8. Uncontrolled intercurrent illness, including ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (excluding insignificant sinus bradycardia and sinus tachycardia) or psychiatric illness/social situations and any other illness that would limit compliance with study requirements and jeopardize the safety of the patient.
* 9. History of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS).
* 10. Pregnant or breast-feeding. Women of childbearing potential must have a pregnancy test performed within 7 days before the enrollment, and a negative result must be documented.
* 11. Previous or concurrent cancer within 3 years prior to treatment start EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer, superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
* 12. Vaccination within 30 days of study enrollment.
* 13. Active bleeding or known hemorrhagic tendency.
* 14. Subjects with unhealed surgical wounds for more than 30 days.
* 15. Being participating any other trials or withdraw within 4 weeks.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Median amount of time subject survives without disease progression following the initiation of treatment | up to 36 months
  The primary endpoint is progression free survival (PFS) after treatment. PFS is defined as the time from first treatment to the date of the first documented tumor progression or death due to any cause.

SECONDARY OUTCOMES:
Number of subjects with treatment related adverse events as assessed by CTCAE v5.0. | Up to 90 days after the last dose of study drugs.
  Establishing the safety profile following the initiation of treatment and grading these toxicities by CTCAE v5.0
The percentage of subjects respond to treatment. | up to 36 months
  Overall response rate is defined as the sum of partial responses and complete responses.
Median amount of times subjects alive after treatment | up tp 36 months
  The median overall survival (OS) time is defined as the time from enrollment to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, PhD, Study Director — Department of Bio-therapeutic, Chinese PLA General Hospital
Locations (1):
- Department of Biotherapeutic, Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No